CLINICAL TRIAL: NCT03342404
Title: A Phase 2, Double-Blind, Randomized, Placebo-Controlled Multicenter Study to Determine the Efficacy and Safety of Luspatercept (ACE-536) Versus Placebo in Adults With Non-Transfusion Dependent Beta (β)-Thalassemia (The BEYOND™ Study)
Brief Title: A Study to Determine the Efficacy and Safety of Luspatercept in Adults With Non Transfusion Dependent Beta (β)-Thalassemia
Acronym: BEYOND
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Collaborators: Acceleron Pharma, Inc., a wholly-owned subsidiary of Merck & Co., Inc., Rahway, NJ USA (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ACE-536-B-THAL-002; U1111-1202-7068 (Registry Identifier: WHO); 2015-003225-33 (EudraCT Number)
Record Dates: First submitted 2017-10-30; First posted 2017-11-17 (Actual); Results first posted 2021-11-18 (Actual); Last update posted 2023-12-20 (Actual); Status verified 2023-11

CONDITIONS: Thalassemia
Keywords: (β)-Thalassemia; Beta-Thalassemia; Phase 2; Luspatercept; ACE-536; Safety; Efficacy; Placebo; Red Blood Cell Transfusions; Erythrocyte transfusion; Hb increase; NTDT
MeSH Terms: conditions — Thalassemia; beta-Thalassemia | interventions — luspatercept; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Luspatercept (ACE-536) plus Best Supportive Care (BSC) (Experimental): Arm Description: Luspatercept, subcutaneous(ly) (SC) once every 21 days
  Interventions: Drug: Luspatercept; Other: Best Supportive Care (BSC)
- Placebo plus Best Supportive Care (BSC) (Placebo Comparator): normal saline solution subcutaneous(ly) (SC) once every 21 days
  Interventions: Other: Placebo; Other: Best Supportive Care (BSC)

INTERVENTIONS:
Drug: Luspatercept — Subjects will start with luspatercept at 1 mg/kg dose level every 3 weeks and can be dose escalated up to 1.25 mg/kg.
  Other Names: ACE-536
  Arms: Luspatercept (ACE-536) plus Best Supportive Care (BSC)
Other: Placebo — Placebo, Subcutaneous, every 21 days
  Other Names: normal saline
  Arms: Placebo plus Best Supportive Care (BSC)
Other: Best Supportive Care (BSC) — Best Supportive Care (BSC)

SUMMARY:
This is a Phase 2, double-blind, randomized, placebo-controlled, multicenter study to determine the efficacy and safety of luspatercept (ACE-536) versus placebo in adults with non-transfusion dependent beta (β)-thalassemia. The study is divided into the Screening Period, Double-blind Treatment Period (DBTP), Open-label Phase (OLP), and Post-Treatment Follow-up Period (PTFP).

It is planned to randomize approximately 150 subjects at a 2:1 ratio of luspatercept versus placebo.

DETAILED DESCRIPTION:
The primary objective is:

- To evaluate the effect of luspatercept (BMS-986346) versus placebo on anemia, as measured by mean hemoglobin concentration in the absence of transfusions over a continuous 12-week interval, from Week 13 to Week 24, compared to baseline.

The secondary objectives are:

* To evaluate the effect of luspatercept versus placebo in anemia-related symptoms in participants with β-thalassemia, as measured by non-transfusion dependent β-thalassemia-patient reported outcome (NTDT-PRO) over continuous 12-week intervals (from Weeks 13 to 24 and from Weeks 37 to 48) compared to baseline.
* To evaluate the effect of luspatercept versus placebo on functional and health-related quality of life (QoL) as measured by Medical Outcomes Study 36-Item Short Form (SF-36) and Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) questionnaires
* To evaluate the long-term effect of luspatercept versus placebo on anemia, as measured by mean hemoglobin concentration in the absence of transfusions over a continuous 12-week interval from Week 37 to Week 48, compared to baseline
* To evaluate the effect of luspatercept versus placebo on iron overload, as measured by liver iron concentration (LIC) and iron chelation therapy (ICT) daily dose
* To evaluate the effect of luspatercept versus placebo on iron overload, as measured by serum ferritin
* To evaluate the duration of erythroid response
* To evaluate the effect of luspatercept versus placebo on physical activity measured by 6-minute walk test (6MWT)

Safety and Pharmacokinetics (PK) Objectives

* To evaluate safety and tolerability of luspatercept, including immunogenicity
* To evaluate population pharmacokinetics (PK) of luspatercept in subjects with β-thalassemia

The exploratory objectives are:

* To evaluate the effect of luspatercept versus placebo on measures of extra-medullary hematopoietic (EMH) masses, bone mineral density, splenomegaly, pulmonary hypertension, and leg ulcers, when present
* To evaluate the effect of luspatercept versus placebo on the β-thalassemia severity as measured by the NTDT severity score system
* To evaluate the effect of luspatercept versus placebo on the β-thalassemia severity as measured by the Morbidity-free Survival parameters
* To examine the relationship of baseline and change in serum Growth Differentiation Factor 11 (GDF11) and other related biomarkers with response to treatment with luspatercept
* To examine the effect of luspatercept on fetal hemoglobin (HbF)
* To examine the effect of luspatercept on Health Resource Utilization (HRU)

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Subjects must be ≥ 18 years of age at the time of signing the informed consent document (ICF).
2. Subject must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
3. Subject is willing and able to adhere to the study visit schedule (eg, not scheduled to receive hematopoietic stem cell transplantation) and other protocol requirements.
4. Subject must have documented diagnosis of β-thalassemia or hemoglobin E/ β-thalassemia. Concomitant alpha globin mutation and/or duplication are allowed.
5. Subject must be non-transfusion dependent, defined as 0 to 5 units of RBCs received during the 24-week period prior to randomization. Note: 1 unit defined for this entry criterion as approximately 200 to 350 mL of transfused packed RBCs.
6. Subject must not be on a regular transfusion program and must be RBC transfusion-free for at least ≥ 8 weeks prior to randomization
7. Subject must have mean baseline hemoglobin ≤ 10 g/dL, based on a minimum of 2 measurements ≥ 1 week apart within 4 weeks prior to randomization; hemoglobin values within 21 days post-transfusion will be excluded.
8. Subject must have performance status: Eastern Cooperative Oncology Group (ECOG) performance score of 0 to 1.
9. A female of childbearing potential (FCBP) for this study is defined as a female who:

1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (ie, has had menses at any time in the preceding 24 consecutive months). A FCBP participating in the study must:

1. Have 2 negative pregnancy tests as verified by the Investigator prior to starting study therapy. She must agree to ongoing pregnancy testing during the course of the study, and after end of study treatment. This applies even if the subject practices true abstinence* from heterosexual contact.
2. Either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis and source documented). If a FCBP engages in sexual activity that may result in a pregnancy, she must agree to use, and be able to comply during the study therapy (including dose interruptions), and for 12 weeks (approximately 5 times the mean terminal half-life of luspatercept based on multiple dose pharmacokinetics [PK] data) after discontinuation of study therapy.

   10. Male subjects must:

a. Practice true abstinence (which must be reviewed on a monthly basis) or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 12 weeks (approximately 5 times the mean terminal half-life of luspatercept based on multiple-dose PK data) following IP discontinuation, even if he has undergone a successful vasectomy

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Any significant medical condition, laboratory abnormality, or psychiatric illness that would prevent the subject from participating in the study.
2. Any condition including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study.
3. Any condition that confounds the ability to interpret data from the study.
4. Diagnosis of hemoglobin S/β-thalassemia or alpha (α)-thalassemia (eg,Hemoglobin H).
5. Active hepatitis C (HCV) infection
6. Deep vein thrombosis (DVT) or stroke requiring medical intervention ≤ 24 weeks prior to randomization.
7. Subjects on chronic anticoagulant therapy are excluded, unless they stopped the treatment at least 28 days prior to randomization. Anticoagulant therapies for prophylaxis and for surgery or high-risk procedures as well as low molecular weight (LMW) heparin for superficial vein thrombosis (SVT) and chronic aspirin are allowed before and during the study.
8. Treatment with another investigational drug or device ≤ 28 days prior to randomization.
9. Prior exposure to sotatercept (ACE-011) or luspatercept (ACE-536).
10. Platelet count > 1000 x 109/L.
11. Subjects on iron chelation therapy (ICT) at the time of ICF signature must have initiated the treatment with ICT at least 24 weeks before the predicted randomization date. ICT can be initiated at any time during treatment and should be used according to the label.
12. Subject had Hydroxyurea and ESA treatment ≤ 24 weeks prior to randomization, and no prior gene therapy.
13. Subject is pregnant or a lactating female.
14. Uncontrolled hypertension. Controlled hypertension for this protocol is considered ≤ Grade 1 according to National Cancer Institute Common Terminology for Adverse Events (NCI CTCAE) version 4.0 (current active minor version).
15. Subject has major organ damage, including:

    1. Liver disease with alanine aminotransferase (ALT) > 3 x upper limit of normal (ULN) or history/evidence of cirrhosis, as well as presence of masses/tumor detected by ultrasound at screening.
    2. Heart disease, heart failure as classified by the New York Heart Association (NYHA) classification 3 or higher, or significant arrhythmia requiring treatment, or recent myocardial infarction (MI) within 6 months of randomization.
    3. Severe lung disease, including pulmonary fibrosis or pulmonary hypertension, ie, ≥G3 NCI CTCAE version 4.0 (current active minor version).
    4. Estimated glomerular filtration rate (eGFR) < 60 ml/min/1.73 m2 (per Modification of Diet in Renal Disease [MDRD] formula).
16. Subject has received chronic systemic glucocorticoids ≤ 12 weeks prior to randomization (physiologic replacement therapy for adrenal insufficiency is allowed).
17. Major surgery ≤ 12 weeks prior to randomization (subjects must have completely recovered from any previous surgery prior to randomization).
18. History of severe allergic or anaphylactic reactions or hypersensitivity to recombinant proteins or excipients in the investigational product (see Investigator Brochure).
19. Subject has received immunosuppressants ≤ 28 days prior to randomization.
20. History or current malignancies (solid tumors and hematological malignancies) unless the subject has been free of the disease (including completion of any active or adjuvant treatment for prior malignancy) for ≥ 5 years. However, subjects with the following history/concurrent conditions are allowed:

    * Basal or squamous cell carcinoma of the skin
    * Carcinoma in situ of the cervix
    * Carcinoma in situ of the breast
    * Incidental histologic finding of prostate cancer (T1a or T1b using the tumor, nodes, metastasis [TNM] clinical staging system)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2018-02-05 (Actual); Primary Completion 2022-11-28 (Actual); Study Completion 2022-11-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeevan Shetty, MD, Study Director — Celgene Corporation
Locations (16):
- United States (4):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - Local Institution - 501, Los Angeles, California
  - Children's Hospital and Research Center at Oakland, Oakland, California
  - Local Institution - 503, Chicago, Illinois
- Greece (2):
  - Local Institution - 102, Athens
  - Local Institution - 101, Athens
- Italy (7):
  - Local Institution - 205, Cagliari
  - Universita degli Studi di Cagliari - ASL8, Cagliari
  - Local Institution - 202, Genoa
  - Local Institution - 201, Milan
  - Local Institution - 203, Naples
  - Local Institution - 206, Napoli
  - Local Institution - 204, Orbassano
- Local Institution - 301, Hazmiyeh, Lebanon
- Local Institution - 401, Bangkok, Thailand
- Local Institution - 601, London Bloomsbury, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Piga A, Perrotta S, Gamberini MR, Voskaridou E, Melpignano A, Filosa A, Caruso V, Pietrangelo A, Longo F, Tartaglione I, Borgna-Pignatti C, Zhang X, Laadem A, Sherman ML, Attie KM. Luspatercept improves hemoglobin levels and blood transfusion requirements in a study of patients with beta-thalassemia. Blood. 2019 Mar 21;133(12):1279-1289. doi: 10.1182/blood-2018-10-879247. Epub 2019 Jan 7. PMID 30617198
- [Derived] Taher AT, Viprakasit V, Kattamis A, Perrotta S, Ricchi P, Porter JB, Coates TD, Forni GL, Musallam KM, Esposito O, Pilot R, Kuo WL, Lai Y, Reverte M, Wei R, Bueno LM, Cappellini MD. Efficacy and safety of luspatercept in non-transfusion-dependent beta-thalassemia: long-term results from the BEYOND study. Blood Adv. 2025 Dec 9;9(23):6108-6119. doi: 10.1182/bloodadvances.2025016554. PMID 40875596
- [Derived] Denton CC, Vodala S, Veluswamy S, Hofstra TC, Coates TD, Wood JC. Splenic iron decreases without change in volume or liver parameters during luspatercept therapy. Blood. 2023 Nov 30;142(22):1932-1934. doi: 10.1182/blood.2023021839. PMID 37704579
- [Derived] Taher AT, Musallam KM, Viprakasit V, Kattamis A, Lord-Bessen J, Yucel A, Guo S, Pelligra C, Shields AL, Shetty JK, Miteva D, Bueno LM, Cappellini MD. Psychometric evaluation of the NTDT-PRO questionnaire for assessing symptoms in patients with non-transfusion-dependent beta-thalassaemia. BMJ Open. 2023 Mar 22;13(3):e066683. doi: 10.1136/bmjopen-2022-066683. PMID 36948565
- [Derived] Taher AT, Cappellini MD, Kattamis A, Voskaridou E, Perrotta S, Piga AG, Filosa A, Porter JB, Coates TD, Forni GL, Thompson AA, Tartaglione I, Musallam KM, Backstrom JT, Esposito O, Giuseppi AC, Kuo WL, Miteva D, Lord-Bessen J, Yucel A, Zinger T, Shetty JK, Viprakasit V; BEYOND Investigators. Luspatercept for the treatment of anaemia in non-transfusion-dependent beta-thalassaemia (BEYOND): a phase 2, randomised, double-blind, multicentre, placebo-controlled trial. Lancet Haematol. 2022 Oct;9(10):e733-e744. doi: 10.1016/S2352-3026(22)00208-3. Epub 2022 Aug 22. PMID 36007538
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.BMSStudyConnect.com

RESULTS

PARTICIPANT FLOW:
Groups:
- Luspatercept: Luspatercept was administered as subcutaneous injection once every 3 weeks (administered on Study Day 1 of each 21-day treatment cycle). The starting dose level was 1.00 mg/kg and could be escalated to 1.25 mg/kg and/or reduced to 0.80, 0.60, and 0.45 mg/kg. Participants were treated for a minimum of 48 weeks.
- Placebo: Placebo (0.9% sodium chloride for injection) was administered as subcutaneous injection once every 3 weeks (administered on Study Day 1 of each 21-day treatment cycle) for a minimum of 48 weeks. Eligible participants entered an open-label phase and started Luspatercept treatment for up to approximately 24 months.
Period: Blinded Treatment Phase
Arm/Group | Luspatercept | Placebo
Started | 96 | 49
Completed | 68 | 18
Not Completed | 28 | 31
Not completed — Withdrawal by Subject | 17 | 10
Not completed — Lack of Efficacy | 2 | 17
Not completed — Adverse Event | 5 | 4
Not completed — Noncompliance with study drug | 1 | 0
Not completed — Other reasons | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Death | 1 | 0
Period: Open-Label Phase
Arm/Group | Luspatercept | Placebo
Started | 0 | 38
Completed | 0 | 27
Not Completed | 0 | 11
Not completed — Lost to Follow-up | 0 | 1
Not completed — Other reasons | 0 | 1
Not completed — Adverse Event | 0 | 3
Not completed — Withdrawal by Subject | 0 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Luspatercept | Placebo | Total
Number analyzed (Participants) | 96 | 49 | 145
Age, Continuous [Mean (Standard Deviation); unit: Years] | 39.3 (13.24) | 41.1 (11.90) | 39.9 (12.79)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 56 | 26 | 82
  Male | 40 | 23 | 63
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 1 | 3
  Not Hispanic or Latino | 94 | 48 | 142
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: Asian | 31 | 13 | 44
  Race: White | 59 | 28 | 87
  Race: Other | 6 | 8 | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Achieving Erythroid Response (Week 13 to Week 24)
Description: Erythroid Response is defined as an increase from baseline ≥1.0 g/dL in mean of hemoglobin values over a continuous 12-week interval from Weeks 13 to 24 of treatment in the absence of transfusions. Baseline hemoglobin (Hb) is the average of 2 or more Hb measurements at least 1 week apart within 4 weeks prior to Dose 1.
Time Frame: From Week 13 to Week 24 of study treatment
Population: All treated participants. Placebo participants are assessed up to crossing over to luspatercept. The luspatercept group does not include placebo participants who crossed over to luspatercept.
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 96 | 49
Percent of Participants | 77.1 [67.4 to 85.0] | 0.0 [0.0 to 7.3]
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Test type: Superiority; Difference in proportions = 77.1, 95% CI 2-sided [63.4 to 87.0] — The difference in proportions (luspatercept - placebo) and 95% CI were estimated from the exact unconditional test
Statistical Analysis 2: Comparison: Luspatercept vs Placebo; Test type: Superiority; Risk Difference (RD) = 77.1, 95% CI 2-sided [68.7 to 85.5] — The common risk difference (luspatercept - placebo) and 95% CI were estimated from the CMH test stratified by baseline Hb category and baseline NTDT-PRO T/W domain score category

2. Secondary Outcome: Mean Change From Baseline in Non-Transfusion Dependent β-thalassemia-Patient Reported Outcome (NTDT-PRO) Tiredness and Weakness (T/W) Domain Score (Week 13 to Week 24)
Description: The NTDT-PRO assesses the severity of anemia-related symptoms with a daily recall of symptoms composed of 6 items: 1. Tiredness (lack of energy) when not doing physical activity 2. Tiredness when doing physical activity 3. Weakness (lack of strength) when not doing physical activity 4. Weakness when doing physical activity 5. Shortness of breath when not doing physical activity 6. Shortness of breath when doing physical activity. The Tiredness/Weakness (T/W) domain score is the average score of items 1 through 4 above. T/W domain score ranges from 0 (best outcome, no tiredness/weakness) to 10 (worst outcome, extreme tiredness/weakness). Weekly T/W Scores are the average of daily scores for that week. The mean of weekly scores over a continuous 12-week period (from Week 13 to Week 24) are compared to the T/W Domain Score at baseline. Baseline is defined as the last value taken on or before the first dose of study drug administered in Week 13.
Time Frame: Baseline and over a continuous 12 week period (from week 13 through week 24)
Population: All treated participants with available measurements at Baseline and from Week 13 to Week 24. Placebo participants are assessed up to crossing over to luspatercept. The luspatercept group does not include placebo participants who crossed over to luspatercept.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 94 | 48
Score on a scale | -0.68 (0.176) | -0.20 (0.240)
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Test type: Superiority; p = 0.0924, ANCOVA; Mean Difference (Net) = -0.48, 95% CI 2-sided [-1.03 to 0.08]

3. Secondary Outcome: Mean Change From Baseline in Hemoglobin Values in the Absence of Transfusion (Week 13 to Week 24)
Description: Mean change from baseline in mean of hemoglobin (Hb) values over a continuous 12-week interval from Week 13 to Week 24 in the absence of transfusions. Baseline was defined as the average of 2 or more Hb measurements at least 1 week apart within 4 weeks before Dose 1 Day 1.
Time Frame: Baseline and over a continuous 12 week period (from week 13 through week 24)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 96 | 47
g/dL | 1.48 (0.078) | 0.07 (0.108)
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Net) = 1.42, 95% CI 2-sided [1.16 to 1.67]

4. Secondary Outcome: Percentage of Participants Achieving Erythroid Response (Week 37 to Week 48)
Description: Erythroid Response is defined as an increase from baseline ≥1.0 g/dL in mean of hemoglobin values over a continuous 12-week interval from Weeks 37 to 48 of treatment in the absence of transfusions. Baseline hemoglobin (Hb) is the average of 2 or more Hb measurements at least 1 week apart within 4 weeks prior to Dose 1.
Time Frame: Assessed over a continuous 12 week period (from week 37 through week 48)
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 96 | 49
Percentage of Participants | 70.8 [60.7 to 79.7] | 2.0 [0.1 to 10.9]
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Mean Difference (Net) = 68.8, 95% CI 2-sided [54.3 to 80.4]

5. Secondary Outcome: Mean Change From Baseline in Mean Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Fatigue Subscale Score (Week 13 to Week 24)
Description: The FACIT-F is a multidimensional, self-report quality of life instrument which includes the Functional Assessment of Cancer Therapy - General (FACT-G) questionnaire (27 items over 4 different domains), and the Fatigue subscale (FS) component (13 items). FACIT-F version 4 has been used for this study. For the Fatigue subscale, each of the 13 items is scored from 0 ("not at all") to 4 ("very much"). The scores from individual items are summed to generated the final FS score, which ranges from 0 (best outcome) to 52 (worst outcome). The questionnaire is completed every other dose, and the mean of FS scores from Week 13 to Week 24 is compared to the FS score at baseline (last score available before start of study treatment). Baseline is defined as the last value taken on or before the first dose of study drug administered in Week 13.
Time Frame: Baseline and over a continuous 12 week period (from week 13 through week 24)
Population: All treated participants with available measurements at Baseline and at least one post-baseline FACIT-F questionnaire completed. Placebo participants are assessed up to crossing over to luspatercept. The luspatercept group does not include placebo participants who crossed over to luspatercept.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 90 | 43
Score on a scale | 1.64 (0.774) | 0.26 (1.066)
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Test type: Superiority; p = 0.2641, ANCOVA; Mean Difference (Net) = 1.39, 95% CI 2-sided [-1.06 to 3.83]

6. Secondary Outcome: Mean Change From Baseline in Non-Transfusion Dependent β-thalassemia-Patient Reported Outcome (NTDT-PRO) Shortness of Breath (SoB) Domain Score (Week 13 to Week 24)
Description: The NTDT-PRO V2.1 assess the severity of anemia-related symptoms associated with NTD β-thalassemia. It is a daily electronic diary with recall of symptoms during the past 24 hours, composed of 6 items: 1. Tiredness (lack of energy) when not doing physical activity 2. Tiredness (lack of energy) when doing physical activity 3. Weakness (lack of strength) when not doing physical activity 4. Weakness (lack of strength) when doing physical activity 5. Shortness of breath when not doing physical activity 6. Shortness of breath when doing physical activity. The Shortness of Breath (SoB) domain score represents the average score of items 5 and 6 above. SoB domain score ranges from 0 (best outcome, no shortness of breath) to 10 (worst outcome, extreme shortness of breath). Weekly SoB Scores represent the average of daily scores for that week. The mean of weekly scores over a continuous 12 week period (from Week 13 to Week 24) are compared to the SoB Domain Score at baseline.
Time Frame: Baseline and over a continuous 12 week period (from week 13 through week 24)
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 94 | 48
Score on a scale | -0.46 (0.168) | 0.02 (0.228)
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Test type: Superiority; p = 0.0721, ANCOVA; Mean Difference (Net) = -0.49, 95% CI 2-sided [-1.02 to 0.04]

7. Secondary Outcome: Mean Change From Baseline in Hemoglobin Values in the Absence of Transfusion (Week 37 to Week 48)
Description: Mean change from baseline in mean of hemoglobin (Hb) values over a continuous 12-week interval from Week 37 to Week 48 in the absence of transfusions. Baseline was defined as the average of 2 or more Hb measurements at least 1 week apart within 4 weeks before Dose 1 Day 1.
Time Frame: Baseline and over a continuous 12 week period (from week 37 through week 48)
Population: All treated participants with available measurements at Baseline and From Week 37 to Week 48. Placebo participants are assessed up to crossing over to luspatercept. The luspatercept group does not include placebo participants who crossed over to luspatercept.
Measure: Least Squares Mean (Standard Error); unit: g/dL
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 91 | 34
g/dL | 1.50 (0.083) | 0.01 (0.130)
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA; Mean Difference (Net) = 1.49, 95% CI 2-sided [1.20 to 1.79]

8. Secondary Outcome: Mean Change From Baseline in Mean Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Fatigue Subscale Score (Week 37 to Week 48)
Description: The FACIT-F is a multidimensional, self-report quality of life instrument which includes the Functional Assessment of Cancer Therapy - General (FACT-G) questionnaire (27 items over 4 different domains), and the Fatigue subscale (FS) component (13 items). FACIT-F version 4 has been used for this study. For the Fatigue subscale, each of the 13 items is scored from 0 ("not at all") to 4 ("very much"). The scores from individual items are summed to generated the final FS score, which ranges from 0 (best outcome) to 52 (worst outcome). The questionnaire is completed every other dose, and the mean of FS scores from Week 37 to Week 48 is compared to the FS score at baseline (last score available before start of study treatment). Baseline is defined as the last value taken on or before the first dose of study drug administered in Week 37.
Time Frame: Baseline and over a continuous 12 week period (from week 37 through week 48)
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 83 | 33
Score on a scale | 2.43 (0.763) | 0.24 (1.150)
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Test type: Superiority; p = 0.0959, ANCOVA; Mean Difference (Net) = 2.19, 95% CI 2-sided [-0.39 to 4.78]

9. Secondary Outcome: Mean Change From Baseline in Non-Transfusion Dependent β-thalassemia-Patient Reported Outcome (NTDT-PRO) Tiredness and Weakness (T/W) Domain Score (Week 37 to Week 48)
Description: NTDT-PRO V2.1 assess the severity of anemia-related symptoms. It's a daily recall of symptoms during the past 24 hours, composed of 6 items: 1. Tiredness (lack of energy) when not doing physical activity 2. Tiredness when doing physical activity 3. Weakness (lack of strength) when not doing physical activity 4. Weakness when doing physical activity 5. Shortness of breath when not doing physical activity 6. Shortness of breath when doing physical activity. The Tiredness/Weakness (T/W) domain score represents the average score of items 1 through 4 above. T/W domain score ranges from 0 (best outcome, no tiredness/weakness) to 10 (worst outcome, extreme tiredness/weakness). Weekly T/W Scores represent the average of daily scores for that week. The mean of weekly scores over a continuous 12-week period (from Week 37 to Week 48) are compared to the T/W Domain Score at baseline. Baseline is defined as the last value taken on or before the first dose of study drug administered in Week 37.
Time Frame: Baseline and over a continuous 12 week period (from week 37 through week 48)
Population: All treated participants with available measurements at Baseline and at Week 37 to Week 48. Placebo participants are assessed up to crossing over to luspatercept. The luspatercept group does not include placebo participants who crossed over to luspatercept.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 72 | 28
Score on a scale | -0.78 (0.229) | 0.01 (0.347)
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Test type: Superiority; p = 0.0510, ANCOVA; Mean Difference (Net) = -0.79, 95% CI 2-sided [-1.58 to 0.00]

10. Secondary Outcome: Mean Change From Baseline in Non-Transfusion Dependent β-thalassemia-Patient Reported Outcome (NTDT-PRO) Shortness of Breath (SoB) Domain Score (Week 37 to Week 48)
Description: NTDT-PRO V2.1 assess the severity of anemia-related symptoms. It is a daily recall of symptoms during the past 24 hours, composed of 6 items: 1. Tiredness (lack of energy) when not doing physical activity 2. Tiredness when doing physical activity 3. Weakness (lack of strength) when not doing physical activity 4. Weakness when doing physical activity 5. Shortness of breath when not doing physical activity 6. Shortness of breath when doing physical activity. The Shortness of Breath (SoB) domain score represents the average score of items 5 and 6 above. SoB domain score ranges from 0 (best outcome, no shortness of breath) to 10 (worst outcome, extreme shortness of breath). Weekly SoB Scores represent the average of daily scores for that week. The mean of weekly scores over a continuous 12-week period (from Week 37 to Week 48) are compared to the SoB Domain Score at baseline. Baseline is defined as the last value taken on or before the first dose of study drug administered in Week 37.
Time Frame: Baseline and over a continuous 12 week period (from week 37 through week 48)
Population: as for outcome 7
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 72 | 28
Score on a scale | -0.59 (0.212) | 0.47 (0.320)
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Test type: Superiority; p = 0.0047, ANCOVA; Mean Difference (Net) = -1.07, 95% CI 2-sided [-1.80 to -0.33]

11. Secondary Outcome: Percentage of Participants With an Increase From Baseline ≥ 3 in Mean Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Fatigue Subscale Score (Week 13 to Week 24)
Description: The FACIT-Fatigue, is a multidimensional, self-report quality of life instrument. It consists of 27 core items, the Functional Assessment of Cancer Therapy - General (FACT-G) questionnaire, which assesses patient function in 4 domains: Physical, Social/Family, Emotional, and Functional well-being, which is further supplemented by a 13-item measure designed to capture cancer-related fatigue, the Fatigue subscale (FS). The items are measured on a response scale with five options (0 = not at all to 4 = very much). Participants completed the questionnaire at screening and every other dose. Baseline is defined as the last value taken on or before the first dose of study drug administered in Week 13. Score is calculated by multiplying the sum of item scores by the n of items in the scale, then divided by n of items answered.
Time Frame: Baseline and over a continuous 12 week period (from week 13 through week 24)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 94 | 47
Percent of Participants | 40.4 [30.4 to 51.0] | 27.7 [15.6 to 42.6]
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Test type: Superiority; p = 0.1359, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 1.8, 95% CI 2-sided [0.8 to 4.0]

12. Secondary Outcome: Percentage of Participants With an Increase From Baseline ≥ 3 in Mean Functional Assessment of Chronic Illness Therapy-Fatigue (FACIT-F) Fatigue Subscale Score (Week 37 to Week 48)
Description: The FACIT-Fatigue, is a multidimensional, self-report quality of life instrument. It consists of 27 core items, the Functional Assessment of Cancer Therapy - General (FACT-G) questionnaire, which assesses patient function in 4 domains: Physical, Social/Family, Emotional, and Functional well-being, which is further supplemented by a 13-item measure designed to capture cancer-related fatigue, the Fatigue subscale (FS). The items are measured on a response scale with five options (0 = not at all to 4 = very much). Participants completed the questionnaire at screening and every other dose. Baseline is defined as the last value taken on or before the first dose of study drug administered in Week 37. Score is calculated by multiplying the sum of item scores by the n of items in the scale, then divided by n of items answered.
Time Frame: Baseline and over a continuous 12 week period (from week 37 through week 48)
Population: as for outcome 5
Measure: Number (95% Confidence Interval); unit: Percent of Participants
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 94 | 47
Percent of Participants | 36.2 [26.5 to 46.7] | 21.3 [10.7 to 35.7]
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Test type: Superiority; p = 0.0657, Cochran-Mantel-Haenszel; Odds Ratio (OR) = 2.3, 95% CI 2-sided [0.9 to 5.4]

13. Secondary Outcome: Mean Change From Baseline in the Physical Component Summary (PCS) and Mental Component Summary (MCS) Scores of the Medical Outcomes Study 36-Item Short Form (SF-36)
Description: The SF-36v2 is a 36-item generic PRO questionnaire used to assess patient-reported outcomes. The SF-36 yields scores for 8 domains of health: Physical Functioning (PF), Role-Physical (RP), Bodily Pain (BP), General Health (GH), Vitality (VT), Social Functioning (SF), Role Emotional (RE), and Mental Health (MH) as well as physical component summary (PCS) and mental component summary (MCS) scores. Scores from each of the 8 domains of health are first normalized based on US general population means, then aggregated and transformed so that the scores from each of the 8 domains of health will contribute differently to the determination of PCS and MCS summary scores. PCS and MCS scores range from 0 to 100, with higher scores indicating a better quality of life. Baseline is defined as the last value taken on or before the first dose of study drug administered.
Time Frame: From baseline to Week 24 and from baseline to Week 48 of study treatment
Population: All treated participants with available measurements at Baseline, at Week 24 and at Week 48. Placebo participants are assessed up to crossing over to luspatercept. The luspatercept group does not include placebo participants who crossed over to luspatercept.
Measure: Least Squares Mean (Standard Error); unit: Score on a scale
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 76 | 37
Score on a scale
  Physical Component Summary (PCS) up to Week 24 | 1.00 (0.499) | -0.38 (0.684)
  Physical Component Summary (PCS) up to Week 48: number analyzed (Participants) | 71 | 30
  Physical Component Summary (PCS) up to Week 48 | 1.23 (0.571) | -0.52 (0.822)
  Mental Component Summary (MCS) up to Week 24 | 0.83 (0.674) | -0.71 (0.947)
  Mental Component Summary (MCS) up to Week 48: number analyzed (Participants) | 71 | 30
  Mental Component Summary (MCS) up to Week 48 | 0.81 (0.784) | -1.89 (1.152)
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Mean change from baseline in SF-36 PCS to Week 24; Test type: Superiority; p = 0.0847, Mixed Models Analysis; Mean Difference (Net) = 1.39, 95% CI 2-sided [-0.19 to 2.96]
Statistical Analysis 2: Comparison: Luspatercept vs Placebo; Mean change from baseline in SF-36 PCS to Week 48; Test type: Superiority; p = 0.0712, Mixed Models Analysis; Mean Difference (Net) = 1.75, 95% CI 2-sided [-0.15 to 3.65]
Statistical Analysis 3: Comparison: Luspatercept vs Placebo; Mean change from baseline in SF-36 MCS to Week 24; Test type: Superiority; p = 0.1633, Mixed Models Analysis; Mean Difference (Net) = 1.54, 95% CI 2-sided [-0.63 to 3.72]
Statistical Analysis 4: Comparison: Luspatercept vs Placebo; Mean change from baseline in SF-36 MCS to Week 48; Test type: Superiority; p = 0.0469, Mixed Models Analysis; Mean Difference (Net) = 2.70, 95% CI 2-sided [0.04 to 5.36]

14. Secondary Outcome: Percentage of Participants With Improvement of Iron Overload
Description: Iron overload was measured by Liver Iron Concentration (LIC) and Iron Chelation Therapy (ICT) daily dose. Improvement is defined as: - For participants with baseline LIC ≥3 mg/g: ≥20% reduction in LIC or ≥ 33% decrease in ICT daily dose - For participants with baseline LIC <3 mg/g: no increase in LIC >1 mg/g and not starting treatment with ICT, or no increase in ICT daily dose ≥ 33% (if on ICT at baseline)
Time Frame: Week 24 and Week 48 of study treatment
Population: as for outcome 1
Measure: Number; unit: Percent of participants
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 96 | 49
Percent of participants
  Week 24 | 44.8 | 49.0
  Week 48 | 34.4 | 49.0
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Percentage of participants with improvement of iron overload (LIC/ICT responders) at Week 24; Test type: Superiority; p = 0.4787, Cochran-Mantel-Haenszel; Mean Difference (Net) = -4.2, 95% CI 2-sided [-21.4 to 13.0]
Statistical Analysis 2: Comparison: Luspatercept vs Placebo; Percentage of participants with improvement of iron overload (LIC/ICT responders) at Week 48; Test type: Superiority; p = 0.0827, Cochran-Mantel-Haenszel; Mean Difference (Net) = -14.6, 95% CI 2-sided [-31.5 to 2.4]

15. Secondary Outcome: Mean Change From Baseline in Serum Ferritin
Description: Baseline mean serum ferritin is calculated during the 24 weeks on or prior to dose 1 day 1. Post-baseline mean serum ferritin is calculated as mean of ferritin values during the last 24 weeks on or prior to the end date of the first 24 week or 48 week treatment
Time Frame: Week 24 and Week 48 of study treatment
Population: All treated participants with available measurements at Baseline and at week 24 or week 48. Placebo participants are assessed up to crossing over to luspatercept. The luspatercept group does not include placebo participants who crossed over to luspatercept.
Measure: Least Squares Mean (Standard Error); unit: ug/L
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 92 | 44
ug/L
  Week 24 | 29.32 (22.949) | 2.18 (32.217)
  Week 48 | 84.94 (23.120) | 71.48 (32.457)
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Mean change from baseline in serum ferritin at Week 24; Test type: Superiority; p = 0.5949, ANCOVA; Mean Difference (Net) = 27.14, 95% CI 2-sided [-46.77 to 101.06]
Statistical Analysis 2: Comparison: Luspatercept vs Placebo; Mean change from baseline in serum ferritin at Week 48; Test type: Superiority; p = 0.3454, ANCOVA; Mean Difference (Net) = 13.46, 95% CI 2-sided [-61.01 to 87.93]

16. Secondary Outcome: Mean Change From Baseline in Liver Iron Concentration (LIC)
Description: LIC was measured by Magnetic Resonance Imaging (MRI). Baseline is defined as the last value on or before the first dose of study drug is administered; Postbaseline is defined as the closest visit at Week 24 or Week 48. Participants with LIC value >43 are not included in the analysis.
Time Frame: Week 24 and Week 48 of study treatment
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: mg/g dry weight
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 87 | 45
mg/g dry weight
  Week 24 | -0.30 (0.125) | -0.21 (0.169)
  Week 48: number analyzed (Participants) | 81 | 40
  Week 48 | -0.34 (0.233) | -1.00 (0.329)
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Mean change from baseline in LIC at Week 24; Test type: Superiority; p = 0.6628, ANCOVA; Mean Difference (Net) = -0.09, 95% CI 2-sided [-0.47 to 0.30]
Statistical Analysis 2: Comparison: Luspatercept vs Placebo; Mean change from baseline in LIC at Week 48; Test type: Superiority; p = 0.0859, ANCOVA; Mean Difference (Net) = 0.66, 95% CI 2-sided [-0.09 to 1.42]

17. Secondary Outcome: Percentage of Participants Who Are Transfusion-Free Over 24 Weeks
Description: Transfusion free is defined as the absence of any transfusion during Week 1-24 of study treatment. Participants who discontinued treatment prior to Week 24 were not considered as transfusion free during Week 1-24.
Time Frame: From first dose to Week 24
Population: as for outcome 1
Measure: Number; unit: Percent of Participants
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 96 | 49
Percent of Participants | 89.6 | 67.3
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Percentage of participants who were transfusion free over 24 weeks; Test type: Superiority; p = 0.0013, Cochran-Mantel-Haenszel; Mean Difference (Net) = 22.2, 95% CI 2-sided [5.0 to 38.6]

18. Secondary Outcome: Percentage of Participants Who Are Transfusion-Free Over 48 Weeks
Description: Transfusion free is defined as the absence of any transfusion during Week 1-48 of study treatment. Participants who discontinued treatment prior to Week 48 were not considered as transfusion free during Week 1-48.
Time Frame: From first dose to Week 48
Population: as for outcome 1
Measure: Number; unit: Percent of Participants
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 96 | 49
Percent of Participants | 82.3 | 44.9
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Percentage of Participants Who are Transfusion-Free Over 48 Weeks; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Mean Difference (Net) = 37.4, 95% CI 2-sided [20.9 to 53.0]

19. Secondary Outcome: Duration of the Mean Hemoglobin Increase From Baseline ≥1.0 g/dL
Description: This outcome measure is the cumulative mean of the duration of hemoglobin response for the ≥ 1.0 g/dL during any 12-week rolling period. Any hemoglobin values within 21 days after a transfusion were excluded from the analysis.
Time Frame: From baseline up to approximately 56 months
Population: All participants with a mean hemoglobin increase ≥1.0 g/dL. Placebo participants are assessed up to crossing over to luspatercept. The luspatercept group does not include placebo participants who crossed over to luspatercept.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 91 | 11
Days | 1136.0 (491.86) | 203.3 (170.82)

20. Secondary Outcome: Mean Change From Baseline in the 6-Minute Walk Test (6MWT) Distance
Description: The 6MWT is typically used to objectively assess functional exercise capacity and response to medical interventions in patients with various moderate to severe diseases. Particiapnts are asked to walk as quickly as possible without running along a 30-meter corridor for six minutes, and the total distance covered during that time is measured. Baseline is defined as the last value on or before the first dose of study drug is administered. Postbaseline is defined as the closest visit at Week 24 or Week 48.
Time Frame: From baseline to Week 24 and from baseline to Week 48 of study treatment
Population: as for outcome 15
Measure: Least Squares Mean (Standard Error); unit: Meters
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 87 | 47
Meters
  24 Weeks | 7.20 (7.017) | -8.96 (9.297)
  48 Weeks: number analyzed (Participants) | 86 | 41
  48 Weeks | 8.82 (5.907) | -3.62 (8.141)
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Mean change from baseline in 6MWT distance at Week 24; Test type: Superiority; p = 0.1466, ANCOVA; Mean Difference (Net) = 16.15, 95% CI 2-sided [-5.73 to 38.04]
Statistical Analysis 2: Comparison: Luspatercept vs Placebo; Mean change from baseline in 6MWT distance at Week 48; Test type: Superiority; p = 0.2011, ANCOVA; Mean Difference (Net) = 12.44, 95% CI 2-sided [-6.72 to 31.59]

21. Secondary Outcome: Percentage of Participants With an Increase From Baseline ≥1.5 g/dL in Mean Hemoglobin Values in the Absence of Transfusion
Description: Percentage of participants who have an increase from baseline ≥1.5 g/dL in mean of hemoglobin (Hb) values over a continuous 12-week interval from Week 13 to Week 24 in the absence of transfusions. Baseline was defined as the average of 2 or more Hb measurements at least 1 week apart within 4 weeks before Dose 1 Day 1.
Time Frame: From Week 13 to Week 24 of study treatment
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Percentage of Participants
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 96 | 49
Percentage of Participants | 52.1 [41.6 to 62.4] | 0.0 [0.0 to 7.3]
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Percentage of Participants with an Increase From Baseline ≥1.5 g/dL in Mean Hemoglobin Values in the Absence of Transfusion; Test type: Superiority; p < 0.0001, Cochran-Mantel-Haenszel; Mean Difference (Net) = 52.1, 95% CI 2-sided [36.2 to 66.2]

22. Secondary Outcome: Percentage of Participants With a Decrease From Baseline ≥ RD (= 1) in the Non-Transfusion Dependent β-thalassemia-Patient Reported Outcome (NTDT-PRO) Tiredness and Weakness (T/W) Domain Score
Description: The responder definition (RD) threshold is the individual participant score change over a predetermined time period that will be interpreted as a treatment benefit. The RD for the NTDT-PRO T/W domain score was defined as ≥ 1-point decrease (ie, RD = -1) from baseline over the time from Week 13 to Week 24 or from Week 37 to Week 48. Participants with missing NTDT-PRO T/W scores at the indicated 12-week period are classified as non-responders in the analysis.
Time Frame: From Week 13 to Week 24 and from Week 37 to Week 48 of study treatment
Population: All treated participants with available measurements at Baseline and at the indicated 12-week periods. Placebo participants are assessed up to crossing over to luspatercept. The luspatercept group does not include placebo participants who crossed over to luspatercept.
Measure: Number (95% Confidence Interval); unit: Percent of participants
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 96 | 49
Percent of participants
  Week 13 to week 24 | 37.5 [27.8 to 48.0] | 28.6 [16.6 to 43.3]
  Week 37 to week 48 | 31.3 [22.2 to 41.5] | 18.4 [8.8 to 32.0]
Statistical Analysis 1: Comparison: Luspatercept vs Placebo; Percentage of Participants With a Decrease From Baseline ≥ RD (= 1) in the Non-Transfusion Dependent β-thalassemia-Patient Reported Outcome (NTDT-PRO) Tiredness and Weakness (T/W) Domain Score Week 13 to Week 24; Test type: Superiority; p = 0.1989, Cochran-Mantel-Haenszel; Mean Difference (Net) = 1.7, 95% CI 2-sided [0.8 to 3.7]
Statistical Analysis 2: Comparison: Luspatercept vs Placebo; Percentage of Participants With a Decrease From Baseline ≥ RD (= 1) in the Non-Transfusion Dependent β-thalassemia-Patient Reported Outcome (NTDT-PRO) Tiredness and Weakness (T/W) Domain Score Week 37 to Week 48; Test type: Superiority; p = 0.0733, Cochran-Mantel-Haenszel; Mean Difference (Net) = 2.1, 95% CI 2-sided [0.9 to 5.0]

23. Secondary Outcome: Number of Participants Experiencing Adverse Events
Description: An Adverse Event (AE) is defined as any new untoward medical occurrence or worsening of a pre-existing medical condition in a clinical investigation participant administered study treatment and that does not necessarily have a causal relationship with this treatment. Adverse events are graded on a scale from 1 to 5, with Grade 1 being mild and asymptomatic; Grade 2 is moderate requiring minimal, local or noninvasive intervention; Grade 3 is severe or medically significant but not immediately life-threatening; Grade 4 events are usually severe enough to require hospitalization; Grade 5 events are fatal.
Time Frame: From first dose to 63 days after last dose (up to approximately 56 months)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 96 | 49
Participants
  Treatment-emergent adverse-event (TEAE) | 96 | 48
  Serious TEAE | 23 | 13
  Treatment-related TEAE | 79 | 18
  Treatment-related Serious TEAE | 4 | 0
  TEAE Leading to Death | 1 | 0
  TEAE Leading to Dose Reduction | 11 | 0
  TEAE Leading to Dose Delay | 47 | 11
  TEAE Leading to Study Drug Discontinuation | 5 | 4
  Treatment-related TEAE Leading to Death | 0 | 0
  Treatment-related TEAE Leading to Dose Reduction | 11 | 0
  Treatment-related TEAE Leading to Dose Delay | 10 | 0
  Treatment-related TEAE Leading to Study Drug Discontinuation | 4 | 0

24. Secondary Outcome: Number of Participants With Anti-drug Antibody (ADA) Positive Test for Luspatercept
Description: Presence of anti-drug (ACE-536/Luspatercept) antibodies was assessed every 24 weeks from serum samples. A participant is counted as 'positive' if there is any positive result captured during the study.
Time Frame: From first dose and up to 2 years following last dose, up to approximately 56 months
Population: All treated participants. Placebo participants are assessed up to crossing over to luspatercept. The luspatercept group does not include placebo who crossed over to luspatercept.
Measure: Count of Participants; unit: Participants
Arm/Group | Luspatercept | Placebo
Number analyzed (Participants) | 96 | 49
Participants | 5 | 3

25. Secondary Outcome: Apparent Clearance (CL/F) of Luspatercept
Description: Apparent Clearance (CL/F) of Luspatercept
Time Frame: Doses 1 to 16: at predose (must be collected before first dose), Dose 2 Day 1, Dose 4 Day 1, Dose 6 Day 1, Dose 8 Day 1, Dose 12 Day 1, Dose 16 Day 1, Dose 6 Day 8, Dose 6 Day 15, and every 6 doses (at Dose 22, 28, etc.), up to approx. 48 months
Population: All treated participants who received the study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/day
Arm/Group | Luspatercept
Number analyzed (Participants) | 96
L/day | 0.458 (33.8)

26. Secondary Outcome: Apparent Volume of Distribution of the Central Compartment (V1/F) of Luspatercept
Description: Apparent Volume of Distribution of the Central Compartment (V1/F) of Luspatercept
Time Frame: as for outcome 25
Population: All treated participants who received the study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Luspatercept
Number analyzed (Participants) | 96
Liters | 7.79 (19.6)

27. Secondary Outcome: Time to Reach Maximum Concentration (Tmax) of Luspatercept
Description: Time to Reach Maximum Concentration (Tmax) of Luspatercept
Time Frame: as for outcome 25
Population: All treated participants who received the study drug.
Measure: Median (Full Range); unit: Days
Arm/Group | Luspatercept
Number analyzed (Participants) | 96
Days | 5.50 [4.33 to 6.42]

28. Secondary Outcome: Maximum Concentration (Cmax) of Luspatercept
Description: Maximum Concentration (Cmax) of Luspatercept
Time Frame: as for outcome 25
Population: All treated participants who received the study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Luspatercept
Number analyzed (Participants) | 96
μg/mL | 5.55 (16.9)

29. Secondary Outcome: Maximum Concentration From Steady State (Cmax,ss) of Luspatercept
Description: Maximum Concentration From Steady State (Cmax,ss) of Luspatercept
Time Frame: as for outcome 25
Population: All treated participants who received the study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μg/mL
Arm/Group | Luspatercept
Number analyzed (Participants) | 96
μg/mL | 8.36 (27.7)

30. Secondary Outcome: Area Under the Curve From Steady State (AUCss) of Luspatercept
Description: Area Under the Curve From Steady State (AUCss) of Luspatercept
Time Frame: as for outcome 25
Population: All treated participants who received the study drug.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: day*μg/mL
Arm/Group | Luspatercept
Number analyzed (Participants) | 96
day*μg/mL | 130 (34.4)

ADVERSE EVENTS:
Time Frame: From first dose to 63 days after last dose (up to approximately 56 months)
Groups:
- Open-Label Placebo-Luspatercept: Open-label phase in which participants switched from placebo and started Luspatercept treatment for up to approximately 24 months.
Arm/Group | Luspatercept | Placebo | Open-Label Placebo-Luspatercept
All-Cause Mortality (participants affected / at risk) | 1/96 | 0/49 | 0/38
Serious Adverse Events (participants affected / at risk) | 23/96 | 13/49 | 3/38
Other Adverse Events (participants affected / at risk) | 96/96 | 48/49 | 38/38
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Luspatercept (N=96) | Placebo (N=49) | Open-Label Placebo-Luspatercept (N=38)
Anaemia (Blood and lymphatic system disorders) | 2 | 0 | 0
Extramedullary haemopoiesis (Blood and lymphatic system disorders) | 1 | 1 | 0
Splenomegaly (Blood and lymphatic system disorders) | 1 | 0 | 0
Cardiac failure acute (Cardiac disorders) | 1 | 0 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 0
Ventricular hypokinesia (Cardiac disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0
Oedema peripheral (General disorders) | 1 | 0 | 0
Bile duct stone (Hepatobiliary disorders) | 1 | 0 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 1
Abscess limb (Infections and infestations) | 0 | 1 | 0
COVID-19 (Infections and infestations) | 2 | 0 | 0
COVID-19 pneumonia (Infections and infestations) | 2 | 1 | 0
Dengue haemorrhagic fever (Infections and infestations) | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 2 | 0
Influenza (Infections and infestations) | 0 | 1 | 0
Pharyngitis (Infections and infestations) | 0 | 1 | 0
Pilonidal disease (Infections and infestations) | 1 | 0 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1 | 0
Septic shock (Infections and infestations) | 1 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 0 | 2 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Pulmonary contusion (Injury, poisoning and procedural complications) | 1 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 5 | 1 | 0
Haemoglobin decreased (Investigations) | 0 | 0 | 1
Diabetes mellitus (Metabolism and nutrition disorders) | 1 | 0 | 0
Hypovolaemia (Metabolism and nutrition disorders) | 1 | 0 | 0
Steroid diabetes (Metabolism and nutrition disorders) | 1 | 0 | 0
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Spinal cord compression (Nervous system disorders) | 1 | 0 | 0
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 0
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 0 | 0 | 1
Proteinuria (Renal and urinary disorders) | 1 | 0 | 0
Renal colic (Renal and urinary disorders) | 0 | 1 | 0
Ovarian cyst ruptured (Reproductive system and breast disorders) | 0 | 1 | 0
Prostatic obstruction (Reproductive system and breast disorders) | 1 | 0 | 0
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Haemothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary arterial hypertension (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Luspatercept (N=96) | Placebo (N=49) | Open-Label Placebo-Luspatercept (N=38)
Extramedullary haemopoiesis (Blood and lymphatic system disorders) | 9 | 2 | 2
Palpitations (Cardiac disorders) | 9 | 6 | 4
Tachycardia (Cardiac disorders) | 6 | 2 | 2
Ear pain (Ear and labyrinth disorders) | 3 | 4 | 0
Vertigo (Ear and labyrinth disorders) | 3 | 3 | 0
Abdominal pain (Gastrointestinal disorders) | 18 | 5 | 4
Abdominal pain upper (Gastrointestinal disorders) | 15 | 3 | 5
Dental caries (Gastrointestinal disorders) | 5 | 2 | 0
Diarrhoea (Gastrointestinal disorders) | 25 | 6 | 5
Dyspepsia (Gastrointestinal disorders) | 18 | 2 | 3
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 5 | 3 | 0
Nausea (Gastrointestinal disorders) | 14 | 6 | 1
Toothache (Gastrointestinal disorders) | 15 | 1 | 0
Vomiting (Gastrointestinal disorders) | 11 | 1 | 1
Asthenia (General disorders) | 19 | 5 | 0
Fatigue (General disorders) | 23 | 10 | 8
Influenza like illness (General disorders) | 25 | 3 | 2
Injection site erythema (General disorders) | 5 | 0 | 3
Malaise (General disorders) | 6 | 1 | 1
Oedema peripheral (General disorders) | 6 | 2 | 1
Pain (General disorders) | 4 | 0 | 2
Pyrexia (General disorders) | 30 | 9 | 11
Biliary colic (Hepatobiliary disorders) | 5 | 0 | 0
Immunisation reaction (Immune system disorders) | 18 | 0 | 5
Bronchitis (Infections and infestations) | 6 | 1 | 1
COVID-19 (Infections and infestations) | 34 | 0 | 15
Gastroenteritis (Infections and infestations) | 12 | 2 | 2
Helicobacter infection (Infections and infestations) | 0 | 0 | 2
Influenza (Infections and infestations) | 15 | 5 | 1
Nasopharyngitis (Infections and infestations) | 7 | 0 | 0
Pharyngitis (Infections and infestations) | 21 | 6 | 1
Rhinitis (Infections and infestations) | 9 | 6 | 0
Sinusitis (Infections and infestations) | 4 | 1 | 2
Tonsillitis (Infections and infestations) | 4 | 6 | 1
Tooth abscess (Infections and infestations) | 6 | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 23 | 11 | 1
Fall (Injury, poisoning and procedural complications) | 2 | 0 | 3
Ligament sprain (Injury, poisoning and procedural complications) | 5 | 0 | 0
Muscle strain (Injury, poisoning and procedural complications) | 5 | 0 | 0
Traumatic fracture (Injury, poisoning and procedural complications) | 6 | 0 | 0
Alanine aminotransferase increased (Investigations) | 6 | 1 | 0
Folate deficiency (Metabolism and nutrition disorders) | 5 | 1 | 0
Hyperuricaemia (Metabolism and nutrition disorders) | 8 | 2 | 1
Iron overload (Metabolism and nutrition disorders) | 14 | 5 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 9 | 4 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 37 | 8 | 11
Back pain (Musculoskeletal and connective tissue disorders) | 38 | 6 | 14
Bone pain (Musculoskeletal and connective tissue disorders) | 42 | 3 | 8
Muscle spasms (Musculoskeletal and connective tissue disorders) | 3 | 1 | 2
Muscular weakness (Musculoskeletal and connective tissue disorders) | 3 | 3 | 1
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 6 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 1 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 16 | 5 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 12 | 2 | 1
Osteoporosis (Musculoskeletal and connective tissue disorders) | 6 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 29 | 5 | 6
Pain in jaw (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3
Spinal pain (Musculoskeletal and connective tissue disorders) | 6 | 1 | 0
Tendonitis (Musculoskeletal and connective tissue disorders) | 5 | 1 | 1
Dizziness (Nervous system disorders) | 19 | 4 | 3
Headache (Nervous system disorders) | 44 | 10 | 10
Migraine (Nervous system disorders) | 9 | 0 | 0
Sciatica (Nervous system disorders) | 5 | 0 | 1
Anxiety (Psychiatric disorders) | 10 | 0 | 1
Insomnia (Psychiatric disorders) | 14 | 1 | 1
Albuminuria (Renal and urinary disorders) | 2 | 0 | 2
Dysuria (Renal and urinary disorders) | 6 | 1 | 0
Renal cyst (Renal and urinary disorders) | 1 | 3 | 0
Dysmenorrhoea (Reproductive system and breast disorders) | 8 | 1 | 1
Menstruation irregular (Reproductive system and breast disorders) | 13 | 3 | 2
Ovarian cyst (Reproductive system and breast disorders) | 3 | 1 | 3
Cough (Respiratory, thoracic and mediastinal disorders) | 24 | 1 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 5 | 0 | 1
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 12 | 1 | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 8 | 2 | 1
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 23 | 6 | 1
Pleuritic pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 2
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 7 | 3 | 0
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 1
Erythema (Skin and subcutaneous tissue disorders) | 7 | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 0 | 2
Skin ulcer (Skin and subcutaneous tissue disorders) | 7 | 1 | 1
Hypertension (Vascular disorders) | 21 | 1 | 7
Prehypertension (Vascular disorders) | 23 | 7 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol-Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single-center publications until after disclosure of the clinical trial's primary publication.

DOCUMENTS (2):
  • Study Protocol (2020-06-12): https://cdn.clinicaltrials.gov/large-docs/04/NCT03342404/Prot_000.pdf
  • Statistical Analysis Plan (2020-11-05): https://cdn.clinicaltrials.gov/large-docs/04/NCT03342404/SAP_001.pdf